CLINICAL TRIAL: NCT02352636
Title: The Experiences for Receiving Auriculotherapy for Osteoarthritis Knee: A Randomised Controlled Feasibility Study.
Brief Title: Auriculotherapy for Osteoarthritis Knee
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: The Hong Kong Polytechnic University (Other)
Responsible Party: Principal Investigator, Lorna Suen, Associate Professor, The Hong Kong Polytechnic University
Allocation: Randomized | Model: Factorial | Masking: Double | Purpose: Treatment
Other Study IDs: G-YBBR
Record Dates: First submitted 2015-01-23; First posted 2015-02-02 (Estimated); Last update posted 2016-08-16 (Estimated); Status verified 2016-08

CONDITIONS: Knee Osteoarthritis
MeSH Terms: conditions — Osteoarthritis, Knee | interventions — Magnetic Field Therapy

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- Treatment arm 1 (Active Comparator): Subjects will receive magnetotherapy (MAT). The magnetic pellets will contain an average of ~200 gauss/pellet magnetic flux densities, with a diameter of 1.76 mm. The experimental object will be applied to the reactive region of each of the six selected acupoints as detected by an acupoint detector. The justifications for selecting these acupoints are described below. To achieve a blinding and placebo effect of the subject, the laser device will be switched to "power off" mode (i.e. deactivated laser) for acupoint "stimulation" prior to the application of MAT. Subjects will be asked to wear a pair of laser protective goggles to "blind" them during therapy administration.
  Interventions: Other: magnetotherapy
- Treatment arm 2 (Active Comparator): Subjects will receive laser auriculotherapy (LAT). A laser device (pointer pulse) will be used in this study. This device has a wavelength of 650 nm, an average output power of 2.5 mW, energy density of 1 minute with 0.54 J/cm2, and a pulse of 10 Hz, which is a common acceptable dosage for clinical use12, 26. This application belongs to a low-energy laser therapy (LLLT), in which the energy level emitted from the device is approximately comparable to a teaching pointer. A 1-minute treatment using the continuous mode of the device will be directly applied to the reactive region of each of the six selected acupoints on the ear. Laser protective goggles will be provided to the subjects and the researchers for eye protection. Similarly, a plaster without magnetic pellets that mimics MAT treatment will be applied on these six acupoints after LAT.
  Interventions: Device: laser auriculotherapy
- Treatment arm 3 (Experimental): Subjects will receive a combined approach using MAT and LAT. LAT will be administered prior to the application of MAT on the selected auricular points, which would be implemented similar to the procedures in treatment arm 1 and 2.
  Interventions: Other: magnetotherapy; Device: laser auriculotherapy
- Placebo arm (Placebo Comparator): Subjects will serve as a placebo control, and will receive LAT at "power off" mode (i.e. deactivated laser) for acupoint "stimulation" before the application of plaster without magnetic pellets that mimic MAT treatment.
  Interventions: Other: Placebo

INTERVENTIONS:
Other: magnetotherapy — The magnetic pellets will contain an average of ~200 gauss/pellet magnetic flux densities, with a diameter of 1.76 mm
  Arms: Treatment arm 1; Treatment arm 3
Device: laser auriculotherapy — A laser device (pointer pulse) will be used in this study. This device has a wavelength of 650 nm, an average output power of 2.5 mW, energy density of 1 minute with 0.54 J/cm2, and a pulse of 10 Hz, which is a common acceptable dosage for clinical use. This application belongs to a low-energy laser therapy (LLLT), in which the energy level emitted from the device is approximately comparable to a teaching pointer.
  Arms: Treatment arm 2; Treatment arm 3
Other: Placebo — Subjects will serve as a placebo control, and will receive LAT at "power off" mode (i.e. deactivated laser) for acupoint "stimulation" before the application of plaster without magnetic pellets that mimic MAT treatment.
  Arms: Placebo arm

SUMMARY:
Osteoarthritis (OA) is the most common form of arthritis in Hong Kong and a prevalent condition in the ageing population. With disease progression, some clients may develop severe pain and profound limitations in ambulation, which may result in morbidity and impaired physical functions. Among the available treatments, pharmacological therapies primarily focus on musculoskeletal pain relief. However, adverse effects, such as gastrointestinal haemorrhage arising from non-steroidal anti-inflammatory drugs have led to an increasing number of concerns regarding the use of these treatments. Other non-invasive complementary methods for osteoarthritic knee (OA knee) should be explored because of the limitations of pharmacological therapy.

Auriculotherapy (AT) is one of the approaches in traditional Chinese medicine (TCM). It is a therapeutic method by which specific points on the auricle are stimulated to treat various disorders of the body. The present study is a four-arm randomised controlled study to determine the effectiveness of AT using magneto-AT (MAT) and/or laser AT (LAT) to improve the conditions of elderly patients suffering from OA knee. The effectiveness of MAT and LAT in terms of alleviating pain, relieving stiffness and promoting a range of motion, and enhancing functional abilities will be determined.

Subjects in 'Treatment arm 1' will receive MAT on specific auricular points on one side of the ear during each treatment session. A deactivated laser will be used to achieve the effect of subject blinding. Subjects in 'Treatment arm 2' will receive LAT using low-energy laser applied to selected acupoints of the ear, and a plaster centred with a portion of Junci Medulla that mimics MAT treatment will also be given. Subjects in 'Treatment arm 3' will receive a combined approach (both MAT and LAT). Subjects in the 'placebo arm' will serve as placebo controls. Six auricular acupoints that are considered to have an effect on the OA knee will be selected. Only one ear at a time will receive treatment. Thus, the ears will be treated alternately. The total treatment period will be four weeks. The experimental objects will be replaced every other day. Therefore, treatment will be performed thrice a week. Subjects will be assessed at baseline up to 3 months after the therapy. This study could advance the knowledge on the complementary approaches than can be used to improve OA knee conditions in the elderly.

DETAILED DESCRIPTION:
Objectives of study

1. To assess the feasibility of AT among elders with OA knee in a future large-scale study, including the use of blinding (subjects and evaluator), acceptance of treatment protocol, follow-up for repetitive testing, estimating effect size and attrition rate.
2. To evaluate the preliminary effect of MAT, LAT or a combined approach among elders with OA knee.
3. To elicit subjects' experiences towards the use of AT in this clinical trial.

Design: This study is a double-blinded randomised controlled trial with a 2 x 2 factorial design, nested with a qualitative study to elicit the experiences of subjects towards the use of AT for OA knee.

Stage I: RCT with factorial design Experimental and control interventions Eligible subjects will be randomly and blindly allocated to one of the four groups, to be decided by a computer-generated randomised table. Restricted randomisation by blocking will be used to ensure approximately similar sample sizes for each group at any time during the trial according to equal proportion rule (1:1:1:1). The random allocation sequence will be managed by a specified research assistant (RA) who is not involved in this trial and is concealed to the assessors.

Treatment arm 1 (MAT & placebo LAT): Subjects will receive MAT. The magnetic pellets will contain an average of ~200 gauss/pellet magnetic flux densities, with a diameter of 1.76 mm. The experimental object will be applied to the reactive region of each of the six selected acupoints as detected by an acupoint detector. The justifications for selecting these acupoints are described below. To achieve a blinding and placebo effect of the subject, the laser device will be switched to "power off" mode (i.e. deactivated laser) for acupoint "stimulation" prior to the application of MAT. Subjects will be asked to wear a pair of laser protective goggles to "blind" them during therapy administration.

Treatment arm 2 (LAT & placebo MAT): Subjects will receive LAT. A laser device (pointer pulse) will be used in this study. This device has a wavelength of 650 nm, an average output power of 2.5 mW, energy density of 1 minute with 0.54 J/cm2, and a pulse of 10 Hz, which is a common acceptable dosage for clinical use. This application belongs to a low-energy laser therapy (LLLT), in which the energy level emitted from the device is approximately comparable to a teaching pointer. A 1-minute treatment using the continuous mode of the device will be directly applied to the reactive region of each of the six selected acupoints on the ear. Laser protective goggles will be provided to the subjects and the researchers for eye protection. Similarly, a plaster without magnetic pellets that mimics MAT treatment will be applied on these six acupoints after LAT.

Treatment arm 3 (Combined MAT & LAT): Subjects will receive a combined approach using MAT and LAT. LAT will be administered prior to the application of MAT on the selected auricular points, which would be implemented similar to the procedures in groups A and B.

Placebo arm: Subjects will serve as a placebo control, and will receive LAT at "power off" mode (i.e. deactivated laser) for acupoint "stimulation" before the application of plaster without magnetic pellets that mimic MAT treatment.

To enhance the blinding effect of the subjects, the following procedures are standardized across the four groups: (1) The auricle of the participant is cleaned using 75% isopropyl alcohol prior to the administration of the therapy; (2) only one ear receives treatment at a time, with both ears treated alternately; (3) all treatment is firstly applied to the right ear in the first visit, followed by the left ear in the second visit, and so on; (4) the experimental objects are replaced every other day, thrice a week (except Sunday) to avoid local irritation of the auricular points under treatment; (5) all subjects will be given an education talk and a booklet on knee OA before the commencement of the study. The total treatment period will last for 4 weeks, with follow up visits at 1-month and 3-month. Therefore the total number of visits for each subject is 15 (i.e. 3 times a week for four weeks, and 2 follow up visits).

Ear zone selection and identification Six auricular acupoints that are thought to have an effect on OA knee are selected, namely, "shenmen", "knee", "spleen", "liver", "kidney" and "subcortex". The Chinese Standard Ear-Acupoints Chart, which is recognised by the World Health Organization, is used to locate the zones. Selection of auricular acupoints is based on traditional Chinese medical theory as well as ideas borrowed from modern medicine.

Participants and settings Subjects 60 years old or above will be recruited from the community centres or day care centres of NGO partners. The therapies will be administered either in the Integrative Health Clinic of the School of Nursing, The Hong Kong Polytechnic University or in the elderly centres, wherever is convenient to the subjects. All therapies will be administered in a room assigned for research purposes. Only the researchers and the client under treatment will be allowed to stay in the room during the therapy. A warning sign on the caution of laser radiation will be put up in a visible place outside the room for other workers or members of the elderly centres.

Inclusion/exclusion criteria The OA condition will be assessed by physical examination based on the clinical criteria of the American College of Rheumatology criteria. The clinical criteria consisted of pain in the knee and any three of the following: (1) aged 50 years of age or over; (2) <=30 minutes of morning stiffness; (3) crepitus on active joint motion; (4) bony tenderness; (5) bony enlargement; or (6) no palpable joint warmth. This classification has been reported to yield 84% specificity and 89% sensitivity for diagnosis of OA knee.

The exclusion criteria were: (1) other connective tissue diseases affecting the knee; (2) knee joint steroid injections within the preceding three months; (3) having a hearing aid or pacemaker in situ (this is to avoid possible interaction between the pacemaker and the magnetic pellets); (4) receiving AT within the preceding three months; (5) suffering from aural injuries or infections; and (6) inability to understand instructions or give consent. The assessment is conducted by a research assistant who will receive intensive coaching on the physical assessment and therapy administration by the research team. Potential subjects will be further assessed by a registered medical practitioner who has over 15 years of clinical experience when the assessment on the OA condition by the RA and the research team is in doubt.

Proposed sample size A total of 96 subjects (24/group) will be recruited in this feasibility study, taking into account of an estimated attrition rate of 20%. The primary outcome of the study, i.e. the pain intensity measured by the Numeric Rating Scale (NRS), is used to determine the effect size of the study.

Ethical considerations A written informed consent will be obtained from every participant after the risks and benefits of the study have been explained to them verbally and in writing. Participation in the study is on a voluntary basis, and all potential participants will be informed and assured that they have the right to refuse or withdraw from the study at any time. Personal information and data will remain confidential and anonymous. Side effects arising from MAT are rare. However, abnormal phenomena such as mild dizziness during or after the procedure or allergic reactions to the skin from the adhesive tape may be possible. Such reactions will be diminished very quickly when the tape is removed, and the frequency of the occurrence of such reverse actions will be monitored closely and recorded. For LAT, the procedure is painless. The subject may sometimes feel a slightly warm feeling on the acupoints under administration when the subjects experienced the "Deqi" feeling which can be seen as a benchmark of effective treatment. Laser protective goggles specific for the wavelength of the laser device will be provided to the subjects and the researchers for eye protection. For the qualitative interview, all interviews will be tape recorded with the permission of the participants. Application for ethical approval from the Human Research Ethics Review Committee, The Hong Kong Polytechnic University, will be applied.

Stage II: Qualitative interviews Semi-structured interviews will be conducted on different group of subjects to elicit a detailed description of the participants' experiences towards the therapy. Purposive sampling will be employed and potential interviewees will be recruited from those who have participated in stage I of the study. Participants from each arm will be recruited. The interview will be conducted in Cantonese and will be tape recorded. The interview guide will serve as a starting point of the interview and an assurance that all relevant topics will be addressed. Open-ended questions, rather than closed-ended or leading questions, will be used to allow the participants to expound on their responses and obtain thick descriptions. Due to the lack of qualitative research on this research topic, the interview questions and probes are not literature based. The interview guide is developed by the first and third investigators based on their clinical experience with the use of AT.

The length of each interview will be moderate and will last for 40 minutes on average. Interviews will be conducted in the participants' homes or at the Integrated Health Clinic (IHC) of the School of Nursing. Two researchers will collect the data: one will conduct the interview, and the other will audio-record the interview and take field notes. Clarification is made by using field notes and probing to ensure the data are not misinterpreted. The interviewer recognized and put aside personal views to minimize subjective bias. Interview will end until data saturation that means no new insight will be generated or no further codes emerged from analysis of interview transcripts.

(b) Qualitative data analyses Interviews conducted in Cantonese will be tape-recorded and transcribed verbatim. A constant comparison method will be used for data analysis not only to describe the phenomenon of interest, but also to develop codes, categories and themes. Related codes will be combined and labeled as categories, with some categories comprising main themes.

Identified scripts will be translated into English by an experienced bilingual translator. The English version of transcript then undergoes backwards translation which will be used for comparing with the original Chinese transcript. The backwards translation can increase the reliability of the English transcript which will be used for content analysis.

ELIGIBILITY:
Inclusion Criteria:

The OA condition will be assessed by physical examination based on the clinical criteria of the American College of Rheumatology criteria. The clinical criteria consisted of pain in the knee and any three of the following:

1. aged 50 years of age or over;
2. <=30 minutes of morning stiffness;
3. crepitus on active joint motion;
4. bony tenderness;
5. bony enlargement; or
6. no palpable joint warmth.

This classification has been reported to yield 84% specificity and 89% sensitivity for diagnosis of OA knee.

Exclusion Criteria:

1. other connective tissue diseases affecting the knee;
2. knee joint steroid injections within the preceding three months;
3. having a hearing aid or pacemaker in situ (this is to avoid possible interaction between the pacemaker and the magnetic pellets);
4. receiving AT within the preceding three months;
5. suffering from aural injuries or infections; and
6. inability to understand instructions or give consent.

The assessment is conducted by a research assistant who will receive intensive coaching on the physical assessment and therapy administration by the research team. Potential subjects will be further assessed by a registered medical practitioner who has over 15 years of clinical experience when the assessment on the OA condition by the RA and the research team is in doubt.

Min Age: 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 44 (Actual)
Dates: Start 2015-01; Primary Completion 2016-06 (Actual); Study Completion 2016-06 (Actual)

PRIMARY OUTCOMES:
Numerical rating scale of pain (NRS) : | collected at baseline up to 3 months after therapy
  According to the OMERACT III conference, which was conducted to establish a core set of outcome measures for future OA trials, the perception of pain has the highest preference among the core set of efficacy domains. Therefore, pain perception using NRS is adopted in this study as a primary outcome. The use of NRS is also considered as a good first choice to evaluate pain perception for most older adults because of its established psychometric properties, increased ability to discriminate pain levels, and common use in clinical practice. The NRS could be administered in written or verbal form, and it involves asking the subject to select a number, from 1 to 10 to the nearest 0.5 interval, to represent their maximal OA induced knee pain in the recent 2 to 3 days.

SECONDARY OUTCOMES:
(2) Western Ontario and McMaster Universities Osteoarthritis Index (WOMAC) | collected at baseline up to 3 months after therapy
  The WOMAC is a disease-specific instrument with 24 items. Physical function is quantified using this scale from 0 (no difficulty) to 96 (extreme difficulty), indicating the level of difficulty associated with overall functional activities caused by knee pain (5 items), stiffness (2 items), and physical function (17 items). Thus, higher scores indicate worse pain, stiffness, and functional limitations. The Chinese WOMAC, which has acceptable psychometric properties (Cronbach's alpha exceeds 0.7 for stiffness and physical function domains; and ICC exceeds 0.7 for all domains), will be adopted in this study.
Standard goniometer | collected at baseline up to 3 months after therapy
  to measure the active and passive range of movement (ROM) of the knees. With the subject in sitting position, active and passive knee extension and flexion ranges will be recorded twice to calculate an average score. To prevent increasing knee joint ROM caused by repeated knee joint measurements, the subject will be allowed to rest for at least 15 minutes between test sessions.
Timed-up-and-go test (TUGT) | collected at baseline up to 3 months after therapy
  TUGT is performed to assess the ambulation status of the subject. The subject will be requested to get up from a chair and walk at a comfortable and safe pace to a destination 3 meters away, turn around, return to the chair, and sit down again. Two trials will be conducted, that is, the practice trial, and the result of the second trial is recorded with a stopwatch, to the nearest second, as the final score. This test is reported to have a high interrater and intrarater reliability (ICC = 0.99), and has demonstrated a good correlation to the Berg Balance Scale, gait speed, and Barthel Index
Subjects' expectations towards therapy | collected at baseline up to 3 months after therapy
  As it is identified in the literature that patient's expectations may influence clinical outcome independently of the treatment itself, therefore a short questionnaire of 8 items is designed to assess patient expectations towards the therapies that they are receiving. Questions include how much they believe that the MAT or LAT have helped them manage their problem, and how much faith they had in complementary therapies, using 10 point scales in most items, with higher the scores indicating higher agreement or satisfaction with each item. These items are adapted from existing literature24,35 and modified for use in this study. A panel of five experts (two registered TCM practitioners, one gerontologist, one nurse specialist, one academic) will be invited to assess the content validity of this questionnaire, and test-retest reliability at a 2-week interval will be determined.

CONTACTS AND LOCATIONS:
Overall Officials: Lorna Suen, MPH, PhD, Principal Investigator — School of Nursing, The Hong Kong Polytechnic University, Hong Kong.
Locations (2):
- Hong Kong (2):
  - Sai Kung District Community Centre, Hong Kong, Hong Kong
  - The Neighbourhood Advice-Action Council, Hong Kong, Hong Kong

REFERENCES:
- [Derived] Suen LK, Yeh CH, Yeung SK. Using auriculotherapy for osteoarthritic knee among elders: a double-blinded randomised feasibility study. BMC Complement Altern Med. 2016 Jul 29;16:257. doi: 10.1186/s12906-016-1242-6. PMID 27473749